CLINICAL TRIAL: NCT04491032
Title: The Effect of Caudal Epidural Injection Volume on Optic Nerve Sheath Diameter and Cerebral Oxygenation in Pediatric Cases
Brief Title: Pediatric Caudal Injection Volume on Optic Nerve Sheath Diameter and Cerebral Oxygenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aybike Onur Gönen (Other)
Collaborators: Pinar Kendigelen (Unknown); Ayse Cigdem Tutuncu (Other); Kaya, Guner, M.D. (Individual); Senol Emre (Unknown); Rahsan Ozcan (Unknown)
Responsible Party: Sponsor-Investigator, Aybike Onur Gönen, Resident in Anesthesiology and Intensive Care, Istanbul University
Organization: Istanbul University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: 72109855-604.01.01-10728
Record Dates: First submitted 2020-07-27; First posted 2020-07-29 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Anesthesia, Caudal; Pediatrics; Elevated Intracranial Pressure
Keywords: optic nerve sheath diameter; cerebral oximetry; caudal epidural anesthesia
MeSH Terms: conditions — Intracranial Hypertension | interventions — Anesthesia, Caudal

STUDY DESIGN:
Intervention Model Description: Patients will receive either a low or high volume of caudal injection.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigator, who will take and record the measurements, will not know about the volume of caudal injection. Another investigator will analyze the ultrasonography images without any knowledge of the patient or the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Volume (Active Comparator): Caudal anesthesia will be performed with 0.8 ml/kg of the local anesthetic solution
  Interventions: Procedure: Caudal anesthesia
- High Volume (Active Comparator): Caudal anesthesia will be performed with 1.25 ml/kg of the local anesthetic solution
  Interventions: Procedure: Caudal anesthesia

INTERVENTIONS:
Procedure: Caudal anesthesia — Caudal epidural injection will be performed after induction of general anesthesia.

SUMMARY:
Caudal anesthesia is a commonly used neuraxial anesthesia method for children. Injection of a certain volume of fluid into the epidural space for cauda anesthesia may push some cerebrospinal fluid towards the head, which may lead to mild increase of pressures inside the head. Such mild changes are compensated well by healthy individuals and no clinical sequel is seen, however at-risk populations may be affected. We aim to see how different amounts of fluid injected into the epidural space may change two clinical parameters affected by intracranial pressure to determine if a lower volume is safer than a higher one.

DETAILED DESCRIPTION:
Caudal epidural injection of local anesthetic solution is a common neuraxial anesthesia technique that provides excellent peri-operative analgesia in children. Unfused sacral hiatus allows for easy and safe access into the epidural space. Anatomically, injection of a certain volume of fluid over the dural sac inside the closed spinal canal can push the cerebrospinal fluid cranially. This push may lead to increased intracranial pressure. We will measure two findings affected by intracranial pressure (optic nerve sheath diameter and cerebral oxygenation) and compare the effects of two different volumes of caudal injections on these measures.

Children with closed fontanelles and scheduled to undergo elective surgery, for which caudal anesthesia is an effective method for peri-operative analgesia, will be recruited for this study. Injection volume will be determined depending on the level of analgesia required for the surgical procedure. Ultrasonographic measurements of optic nerve sheath diameter and near-infrared spectrometry measurement of cerebral oxygenation will be taken before and after caudal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* ASA class 1 or 2
* Scheduled for elective surgery suitable for caudal anesthesia
* Parental/guardian consent for caudal anesthesia and measurements obtained
* Closed fontanelles

Exclusion Criteria:

* Open fontanelle
* Parental/guardian refusal
* Previous intracranial or ocular pathology
* Coagulapathies
* Variations in gross and ultrasonographic sacral anatomy
* Block performence to end of surgery expected to last less than 30 minutes
* Block volumes more than 30ml needed
* Laparoscopic surgery
* Need for long term analgesia with epidural catheter

Ages: 12 Months to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Change in optic nerve sheath diameter | From before caudal injection to immediately, 10 min, 20 min and 30 min after.
  Difference in the percentage change of ultrasonographic measurement of optic nerve sheath diameter between groups
Change in cerebral oxygenation | From before caudal injection to immediately, 10 min, 20 min and 30 min after.
  Difference in the change in near-infrared spectrometry measurement of cerebral oxygenation between the groups

SECONDARY OUTCOMES:
Variation in optic nerve sheath diameter | From before caudal injection to immediately, 10 min, 20 min and 30 min after.
  Difference in the percentage change of ultrasonographic measurement of optic nerve sheath diameter in each group
Variation in cerebral oxygenation | From before caudal injection to immediately, 10 min, 20 min and 30 min after.
  Difference in the change in near-infrared spectrometry measurement of cerebral oxygenation in each group

OTHER OUTCOMES:
Changes in hemodynamic and respiratory parameters | From before caudal injection to immediately, 10 min, 20 min and 30 min after.
  Mean arterial pressure, heart rate, end-tidal carbondioxide pressure, peak inspiratory pressure, peripheral oxygen saturation, oxygen fraction of inhaled gas

CONTACTS AND LOCATIONS:
Overall Officials: Aybike Onur Gönen, MD, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No formal plans to share IPD is made

REFERENCES:
- [Derived] Gonen AO, Kaya G, Tutuncu AC, Ozcan R, Emre S, Kendigelen P. Effect of paediatric caudal injection volume on optic nerve sheath diameter and regional cerebral oximetry: A randomised trial. Eur J Anaesthesiol. 2023 Jul 1;40(7):465-471. doi: 10.1097/EJA.0000000000001819. Epub 2023 Mar 20. PMID 36938985